CLINICAL TRIAL: NCT03883698
Title: Pharmacokinetics of Low-dose Sofosbuvir in Dialysis-dependent Patients With Hepatitis C Virus Infection
Brief Title: Safety of Sofosbuvir in People With Advanced Kidney Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-167-IMP-107; CTRI/2019/03/018011 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Kidney Failure, Chronic; Hepatitis C
MeSH Terms: conditions — Kidney Failure, Chronic; Hepatitis C | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Intervention Model Description: This is a three arm, case control study aimed at studying the pharmacokinetics of sofosbuvir and its major metabolite (GS-331007) in people with estimated GFR (eGFR) <30 ml/min. Two arms will include participants with advanced renal failure with eGFR below 30 ml/min and third arm will include participants with normal eGFR. Participants with eGFR <30 ml/min will receive sofosbuvir in doses of either 400mg on alternate days or 200mg daily. The participants with normal eGFR will receive the standard of care, i.e, 400mg of sofosbuvir daily
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESRD, alternate day dose (Experimental): Participants with end stage renal disease (eGFR <30 ml/min) and hepatitis C virus active infection and treated with sofosbuvir 400 mg on alternate days. Total duration of treatment will be 12 weeks
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir 60 mg
- ESRD, daily dose (Experimental): Participants with end stage renal disease (eGFR <30 ml/min) and hepatitis C virus active infection and treated with sofosbuvir 200 mg daily doses. The total duration of treatment will be 12 weeks
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir 60 mg
- Control (Active Comparator): Participants with normal eGFR and hepatitis C virus infection and treated with sofosbuvir 400 mg daily dose. The total duration of treatment will be 12 weeks
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir 60 mg

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir is the backbone of the most of the currently used anti-HCV treatment regimens
Drug: Daclatasvir 60 mg — Daclatasvir, in combination with sofosbuvir, is approved for the treatment of hepatitis C virus infection in absence of liver cirrhosis

SUMMARY:
Infection with hepatitis C virus (HCV), a hepatotropic RNA virus, is often chronic, and causes liver cirrhosis and liver cancer. The virus is transmitted through parenteral exposure. This infection is particularly common in those on maintenance hemodialysis.

Sofosbuvir, an inhibitor of HCV RNA-dependent RNA polymerase, forms the backbone of DAA-based anti-HCV treatment regimens. In pre-clinical pharmacokinetic studies, administration of the usual 400 mg daily dose to in presence of advanced kidney failure (estimated glomerular filtration rate [eGFR] of <30 ml/min) showed that serum levels of the sofosbuvir and GS-331007, the primary metabolite of sofosbuvir, were elevated by several folds. Hence, sofosbuvir is not approved for use in people on maintenance hemodialysis.

The newer DAAs (e.g. grazoprevir/elbasvir combination), which have been approved for use in people with eGFR <30 ml/min, are very costly and are not available in Asian countries including India. Hence, as a rescue measures, several physicians, including our group, have tried half-daily dose (i.e, 200 mg daily or 400mg on alternate days) of sofosbuvir and 60 mg daclatasvir in dialysis-dependent people, with good results in terms of both safety and efficacy. In fact, the use of this empirical 200 mg daily dose schedule has become common in clinical practice. However, this use is not based on any pharmacokinetic data.

Hence, it is proposed to study the pharmacokinetics of low-dose (200 mg daily or 400 mg alternate day) of sofosbuvir and GS-331007 metabolite in people with eGFR <30/min and active HCV infection.

DETAILED DESCRIPTION:
Study design Three arms, observational, pharmacokinetic study

Study duration Two years (March 2019-February 2020)

Study participants Two groups of participants will be included (i) People without chronic kidney disease, i.e, normal eGFR and infected with HCV infection (ii) People with chronic kidney disease and eGFR <30 ml/min and infected with HCV infection

We will include a total of thirty participants with ten in each of the three groups: Group A (ESRD, alternate day dose), Group B (ESRD, daily dose) and Group C (normal eGFR)

Drug schedule Participants with eGFR <30 ml/min: will be given daclatasvir 60 mg once daily along with either sofosbuvir (200 mg) daily once or sofosbuvir 400mg once every alternate day Participants with normal renal function will be treated with sofosbuvir 400mg and daclatasvir 60 mg once daily.

The treatment duration will be 12 weeks for alll there three study groups.

Dialysis schedule A four to five hour hemodialysis sessions will be provided twice in a week

Plan for pharmacokinetic study (i) Molecules: Sofosbuvir and GS331007 (ii) Method: Liquid chromatography-tandem mass spectrometry (iii) Specimen collection (~2 ml each time) will be done as follows: Hour '0', 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24 [Day 1]; hour 36 [Day 2]; hour 84 [Day 4], and hour 156 [Day 7].

Sample Collection, Transport and Storage Soon after sample collection, serum will be separated by centrifugation at 4000×g for 10 min at 4°C and separated serum will stored at -80°C till analysis. Analysis will be done using validated bioanalytical method at CSIR-CDRI, Lucknow.

Inactivation of hepatitis C virus in the stored sample HCV inactivation will be done by heat treatment. Before heat treatment, water bath chamber will be cleaned, filled with fresh RO water and temperature calibration will be checked for accuracy. The specimens will be heated at 60 C for 10 minutes or 65 C for 5 minutes to inactivate the virus. Immediately after heat treatment, the specimens will be put in crushed ice to stop the heat effect. The specimens will be transported in frozen condition for analysis.

Sample preparation:

The sample preparation consists of the simple liquid-liquid extraction and/or protein precipitation.

Liquid chromatography-mass spectroscopy HPLC system consisting of Shimadzu UFLC system consisting of LC-20AD binary pumps and SIL-HTc autosampler (Shimadzu Corporation, Kyoto, Japan) will be used to inject 10 µL aliquots of the processed samples on a C18 column (4.6 mm × 50 mm, 5.0 µm). The separation will be achieved by running the mobile phase in isocratic mode containing acetonitrile and 10mM ammonium acetate buffer in suitable ratio (%v/v) at a flow rate capable of sufficient resolution to be optimized during method development and validation. The mobile phase will be duly filtered through 0.22 µm filter and degassed ultrasonically before use. Mass spectrometric detection will be performed on an API 5500 Q Trap mass spectrometer (Applied Biosystems, MDS Sciex Toronto, Canada) equipped with an API electron spray ionization (ESI) source. The ion spray voltage will be set at 5500 V. The instrument related parameters viz., nebulizer gas, curtain gas, auxiliary gas and collision gas and coompound related parameters viz., declustering potential (DP), collision energy (CE), entrance potential (EP) and collision cell exit potential (CXP) respectively will be optimized before validating the method . Zero air will be used as source gas while nitrogen will be used as both curtain and collision gas. The mass spectrometer will be operated at ESI positive as well as ESI negative ion mode and detection of the ions will be performed in the multiple reaction monitoring (MRM) mode monitering the transitions of the analytes. Quadrupole 1 and quadrupole 3 will be maintained at unit resolution and dwell time will be set at 200 ms. Analyst 1.6 software (version 1.6, Built 3773; AB Sciex, Toronto, Canada) will be used for data acquisition and quantitation.

Pharmacokinetic parameters estimation The pharmacokinetic parameters will be estimated using WinNonlin software either through compartment/non-compartment modeling.

ELIGIBILITY:
Inclusion Criteria:

* Participants with:

  * hepatitis C virus infection with detectable HCV RNA in blood
  * naïve to direct acting antiviral drugs based anti-HCV treatment

Exclusion Criteria:

* Hepatitis B virus co-infection
* Human immunodeficiency virus co-infection
* Clinical evidence of cirrhosis or portal hypertension such as ascites, esophageal or gastric varices on esophago-gastro-duodenoscopy, liver stiffness more than 15 KPa as measured with transient elastography or history of hepatic encephalopathy.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics study | At hour (from the time of drug administration) '0', 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24 on Day 1; hour 36 on Day 2; at hour 84 on Day 4; and at hour 156 on Day 7
  To study the Maximum Plasma Concentration [Cmax] of sofosbuvir and its metabolite (GS-331007) in participants with eGFR below 30 ml/min who are treated with low-dose of sofosbuvir and compare it with that in people with normal eGFR.
Pharmacokinetics study | At hour (from the time of drug administration) '0', 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24 on Day 1; hour 36 on Day 2; at hour 84 on Day 4; and at hour 156 on Day 7
  To study the Area Under the Curve [AUC] of sofosbuvir and its metabolite (GS-331007) in participants with eGFR below 30 ml/min who are treated with low-dose of sofosbuvir and compare it with that in people with normal eGFR.
Pharmacokinetics study | At hour (from the time of drug administration) '0', 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24 on Day 1; hour 36 on Day 2; at hour 84 on Day 4; and at hour 156 on Day 7
  To study the Terminal Half Life [t1/2] of sofosbuvir and its metabolite (GS-331007) in participants with eGFR below 30 ml/min who are treated with low-dose of sofosbuvir and compare it with that in people with normal eGFR.

SECONDARY OUTCOMES:
Clinical response | 12 weeks after stopping anti-HCV treatment
  Proportion of participants with sustained virologic response at 12 weeks [SVR12] after discontinuation of anti-HCV treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amit Goel, DM, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGI)
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided
As of now, our group has not decided about sharing the IPD with other researchers in a publicly available platform. Though, if needed, we could try to share the needed information if our institute's ethic committee permits for the same.

REFERENCES:
- [Background] Kirby BJ, Symonds WT, Kearney BP, Mathias AA. Pharmacokinetic, Pharmacodynamic, and Drug-Interaction Profile of the Hepatitis C Virus NS5B Polymerase Inhibitor Sofosbuvir. Clin Pharmacokinet. 2015 Jul;54(7):677-90. doi: 10.1007/s40262-015-0261-7. PMID 25822283
- [Background] European Association for the Study of the Liver. EASL Recommendations on Treatment of Hepatitis C 2018. J Hepatol. 2018 Aug;69(2):461-511. doi: 10.1016/j.jhep.2018.03.026. Epub 2018 Apr 9. No abstract available. PMID 29650333
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Hepatitis C Work Group. KDIGO 2018 Clinical Practice Guideline for the Prevention, Diagnosis, Evaluation, and Treatment of Hepatitis C in Chronic Kidney Disease. Kidney Int Suppl (2011). 2018 Oct;8(3):91-165. doi: 10.1016/j.kisu.2018.06.001. Epub 2018 Sep 19. No abstract available. PMID 30675443
- [Background] Goel A, Bhadauria DS, Kaul A, Verma P, Mehrotra M, Gupta A, Sharma RK, Rai P, Aggarwal R. Daclatasvir and reduced-dose sofosbuvir: An effective and pangenotypic treatment for hepatitis C in patients with estimated glomerular filtration rate <30 mL/min. Nephrology (Carlton). 2019 Mar;24(3):316-321. doi: 10.1111/nep.13222. PMID 29327401